CLINICAL TRIAL: NCT00892541
Title: Investigation of the Potential Effects of Trimethoprim on the Pharmacokinetics of ER OROS Paliperidone in Healthy Male Subjects
Brief Title: A Study of the Potential Effects of Trimethoprim on the Pharmacokinetics of ER OROS Paliperidone
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: CR004150
Record Dates: First submitted 2008-11-20; First posted 2009-05-04 (Estimated); Last update posted 2011-06-08 (Estimated); Status verified 2010-03

CONDITIONS: Schizophrenia
Keywords: Schizophrenia; Mood disorders; Antipsychotic drugs; Renal secretion; ER OROS paliperidone
MeSH Terms: conditions — Schizophrenia; Mood Disorders

INTERVENTIONS:
Drug: ER OROS paliperidone

SUMMARY:
The purpose of this study is to evaluate the effects of an organic cation transporter inhibitor, trimethoprim, on the pharmacokinetics of orally administered ER OROS paliperidone and to assess the safety and tolerability of the treatments in healthy male volunteers.

DETAILED DESCRIPTION:
This study was designed as a single center, open-label, randomized, 2 treatment period crossover study in healthy male volunteers. The study consists of a screening period (within 21 days before the first study drug administration) before randomization; an open-label treatment phase consisting of 2 periods during which subjects will receive a single oral dose of ER OROS paliperidone alone (Treatment A) or in combination with 200 mg trimethoprim twice daily (Treatment B); and end-of-study evaluations upon completion of all the study procedures in Period 2 or early withdrawal. The pharmacokinetic blood and urine samples will be collected over a 96 hour period after ER OROS paliperidone administration. Successive ER OROS paliperidone administrations will be separated by at least 14 days. Given that the main elimination route of paliperidone is renal clearance and about half of this is through active secretion in the renal tubule, competition for this route of elimination can occur when other actively secreted drugs are coadministered. Therefore, the possible influence on the renal excretion of paliperidone will be investigated when a competitor for active renal secretion, trimethoprim, is coadministered. Safety and tolerability will be monitored throughout the study. Treatment A: a single oral dose of 6 mg ER OROS paliperidone on Day 1; Treatment B: a 200 mg trimethoprim tablet twice daily from Day 1 to Day 8 and a single oral dose of 6 mg ER OROS paliperidone on Day 5.

ELIGIBILITY:
Inclusion Criteria:

* Male, aged 18 to 55 years, inclusive
* Volunteers must have signed an informed consent document indicating that they understand the purpose of and procedures required for the study and are willing to participate in the study
* Body Mass Index (BMI, weight [kg]/height [m²]) range of 18 to 28 kg/m², inclusive
* Normotensive with supine (5 minutes) blood pressure between the range of 100 to 140 mmHg systolic, inclusive, and 60 to 90 mmHg diastolic, inclusive
* Healthy on the basis of a prestudy physical examination, medical history, ECG, and the laboratory results of serum chemistry, hematology and urinalysis performed within 21 days before the first dose. If the results of the serum chemistry, hematology or urinalysis testing are not within the laboratory's reference ranges the subject can be included only if the investigator judges that the deviations are not clinically significant
* Creatinine clearance value greater than or equal to 80 mL/min
* Signed an informed consent for genetic testing, indicating whether the volunteer does or does not wish to participate in the genetic part of the study.

Exclusion Criteria:

* Drug allergy to risperidone, paliperidone, trimethoprim, any of its excipients or history of hypersensitivity to heparin, in case a heparin lock will be used
* Past or current history of folic acid deficiency or megaloblastic anemia
* Recent history of alcohol or substance abuse or dependence or a positive test result for the urine drug screen at screening
* Relevant history or presence of any cardiovascular (including myocardial infarct or cardiac arrhythmia), respiratory, neurological (including seizures, cerebrovascular disorders), psychiatric, renal, hepatic, gastrointestinal (including surgeries, severe gastrointestinal narrowing, and malabsorption problems), endocrinal, hematological or immunological disease. History of any cancer, with the exception of basal cell carcinomas
* At screening, has a decrease of >20 mmHg in systolic blood pressure or a decrease of >10 mmHg in diastolic blood pressure after standing for at least 2 minutes that is not associated with an increase of >15 beats per minute (bpm) in heart rate
* Bradycardia (heart rate <45 bpm) as determined by screening ECG
* A positive result for any of the tests for hepatitis B, C, and human immunodeficiency virus (HIV).

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 30 (Actual)
Dates: Start 2004-10; Study Completion 2004-11 (Actual)

PRIMARY OUTCOMES:
To evaluate the effects of an organic cation transporter inhibitor, trimethoprim, on the pharmacokinetics of orally administered ER OROS paliperidone

SECONDARY OUTCOMES:
To evaluate the safety and tolerability of the treatments in healthy male volunteers

CONTACTS AND LOCATIONS:
Overall Officials: Johnson & Johnson Pharmaceutical Research & Development, L.L. C. Clinical Trial, Study Director — Johnson & Johnson Pharmaceutical Research & Development, L.L.C.

REFERENCES:
- See also: A study of the potential effects of trimethoprim on the pharmacokinetics of ER OROS paliperidone — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=557&filename=CR004150_CSR.pdf